CLINICAL TRIAL: NCT03961321
Title: SMART (Stereotactic MR-guided Adaptive Radiation Therapy) for Localized Prostate Cancer; a Phase II Study
Brief Title: Stereotactic MR-guided Adaptive Radiation Therapy for Localized Prostate Cancer
Acronym: SMART
Status: Completed | Type: Observational
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, Anna Bruynzeel, Principal Investigator, Amsterdam UMC, location VUmc
Other Study IDs: NL5728902916
Record Dates: First submitted 2019-05-15; First posted 2019-05-23 (Actual); Last update posted 2019-05-23 (Actual); Status verified 2019-05

CONDITIONS: Prostatic Neoplasms
Keywords: SMART; Prostate cancer; SBRT; MRgRT; Toxicity
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: stereotactic mr guided adaptive radiotherapy — Study patients will be treated with an online MR-guided hypofractionated course of radiotherapy in 5 fractions of 7.25 Gy per fraction delivered on the prostate with a simultaneous integrated sparing (SIS) of the urethra with a dose of 32.5 Gy in 5 fractions (6.5 Gy per fraction).

SUMMARY:
Rationale: This prospective study investigates the outcomes of daily online stereotactic MR-guided adaptive radiation therapy (SMART) in patients with localized prostate cancer (cT1c-T3bN0M0). Visualization of the prostate, rectum and bladder prior to and during radiation delivery can be used to deliver "gated" treatment (beam-on only when the prostate is in the predetermined position) using small uncertainty margins. The novel MRIdian treatment delivery system (ViewRay, USA), which will be used for this study, allows for the immediate generation of an optimal radiotherapy plan based on the current anatomy of the prostate and surrounding normal organs prior to each fraction. These major advances will (i.e. dosimetrically) allow for an optimisation of normal tissue radiation doses, which should theoretically decrease toxicity to surrounding organs such as the rectum or bladder. Another advantage of this approach is that online MR-based prostate imaging does not rely on implanted gold markers, avoiding an invasive procedure to insert such markers. If proven feasible, this approach could set a new standard of care for patients with localized prostate cancer.

The main goal of this phase II study of SMART for prostate cancer is to evaluate the early and early-delayed toxicity, i.e. within the first year after treatment. An established 5-fraction hypofractionated radiation scheme will be used in this trial.

Main outcome parameters will include gastro-intestinal, genitourinary and sexual symptoms, which will be monitored at fixed time points using CTCAE criteria. In addition, patient-reported outcomes will be evaluated using EORTC-QOL questionnaires.

Objective: To investigate the early and early-delayed toxicity profile of SMART in patients with localized prostate cancer.

Study design:phase II observational study Study population: 100 consecutive patients with localized prostate cancer (cT1c-T3bN0M0).

Study intervention: Study patients will be treated with an online MR-guided hypofractionated course of radiotherapy in 5 fractions of 7.25 Gy per fraction delivered on the prostate with a simultaneous integrated sparing of the urethra with a dose of 32.5 Gy in 5 fractions Main study parameters: Early and early-delayed toxicity (CTCAE v. 4.0); (IPSS) and Qol C30 PR25. Secondary endpoint will be the offline evaluation of the dosimetric benefit of SMART by comparing cumulative doses to organs at risk.

DETAILED DESCRIPTION:
Rationale: This prospective study investigates the outcomes of daily online stereotactic MR-guided adaptive radiation therapy (SMART) in patients with localized prostate cancer (cT1c-T3bN0M0). Visualization of the prostate, rectum and bladder prior to and during radiation delivery can be used to deliver "gated" treatment (beam-on only when the prostate is in the predetermined position) using small uncertainty margins. The novel MRIdian treatment delivery system (ViewRay, USA), which will be used for this study, allows for the immediate generation of an optimal radiotherapy plan based on the current anatomy of the prostate and surrounding normal organs prior to each fraction. These major advances will (i.e. dosimetrically) allow for an optimisation of normal tissue radiation doses, which should theoretically decrease toxicity to surrounding organs such as the rectum or bladder. Another advantage of this approach is that online MR-based prostate imaging does not rely on implanted gold markers, avoiding an invasive procedure to insert such markers. If proven feasible, this approach could set a new standard of care for patients with localized prostate cancer.

The main goal of this phase II study of SMART for prostate cancer is to evaluate the early and early-delayed toxicity, i.e. within the first year after treatment. An established 5-fraction hypofractionated radiation scheme will be used in this trial. At VUmc, experience with this scheme has been obtained as a result of participation in a recently concluded multicenter randomized phase II trial [METc NL4181402912; 20012/398]. Main outcome parameters will include gastro-intestinal- (GI), genitourinary- (GU) and sexual symptoms, which will be monitored at fixed time points using CTCAE criteria. In addition, patient-reported outcomes will be evaluated using EORTC-QOL questionnaires.

Objective: To investigate the early and early-delayed toxicity profile of SMART in patients with localized prostate cancer.

Study design: A phase II observational study Study population: 100 consecutive patients with localized prostate cancer (cT1c-T3bN0M0).

Study intervention: Study patients will be treated with an online MR-guided hypofractionated course of radiotherapy in 5 fractions of 7.25 Gy per fraction delivered on the prostate with a simultaneous integrated sparing (SIS) of the urethra with a dose of 32.5 Gy in 5 fractions (6.5 Gy per fraction). This stereotactic radiation scheme was also used in [METc NL4181402912; 20012/398].

Main study parameters: Early and early-delayed toxicity (CTCAE v. 4.0); prostate specific symptom score (IPSS) and Qol (EORTC-QoL C30 & QLQ Prostate Cancer module (QLQ-PR25)). Secondary endpoint will be the offline evaluation of the dosimetric benefit of SMART by comparing cumulative doses to organs at risk.

Nature, extent of the burden and risks associated with participation, benefit and group relatedness: This novel SMART approach could set a new standard of care for patients with localized prostate cancer by limiting radiation doses to surrounding normal organs and thereby potentially radiation-induced toxicity. Also, implantation of gold markers would become unnecessary using MR-guided "gated" radiotherapy. Disadvantages for patients include the need to be positioned within the MRI bore during radiation delivery, and a prolonged time per treatment fraction (estimated at 30 minutes per fraction), which has to be weighed against the use of a total of only five fractions. As the radiation fractionation scheme that is used in this study has been evaluated in prior trials, no further patient-related risks are anticipated.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 years or older
* WHO performance score 0-2
* Biopsy proven adenocarcinoma of the prostate
* Gleason ≥ 6
* Prostate volume ≤ 90 cc on TRUS
* T-stage: cT1c-T3b (on MRI and/or endorectal ultrasound)
* All patients should be able to undergo MRI scans
* No evidence of lymph node or distant metastases on radiological staging
* The multidisciplinary team advised external beam radiotherapy treatment
* IPSS (International Prostate Symptoms Score) ≤19
* Previous TURP is allowed provided there is at least 8 weeks interval with radiotherapy
* The administration of concomitant hormonal therapy is allowed
* Ability to provide written informed consent.

Exclusion Criteria:

* Previous irradiation in the pelvic region
* Contra-indications for MRI

  * As no safety data for 0.35 Tesla MRI scanners are available on electronic devices such as pacemakers or implanted defibrillators, deep brain stimulators, cochlear implants, this constitutes an absolute contraindication for this study, even for devices that have been considered safe for MRI scans with higher magnetic field strengths.
  * Patients who have a metallic foreign body in their eye, or who have an aneurysm clip in their brain, cannot have an MRI scan since the magnetic field may dislodge the metal
  * Patients with severe claustrophobia may not be able to tolerate an MRI scan
  * Patients with a hip prosthesis will not be eligible for the MRI scan

Min Age: 18 Years | Sex: Male
Age Groups: Adult, Older Adult
Gender Based: Yes — prostate cancer
Study Population: Patients with localized prostate cancer with a clinical stage T1-3b, with a maximal volume of 90 cc on transrectal ultrasound (TRUS) and no suspicious lymph nodes observed on either a diagnostic MRI or CT scan and no signs of distant metastases on radiological staging are eligible. All patients will be discussed in the multidisciplinary board (MDO) with an urologist, medical oncologist, radiologist, pathologist and a radiation oncologist, all specialized in the treatment of prostate cancer. If the MDO treatment advise comprises external beam radiotherapy, patient eligibility for the study will be assessed, and the treating radiation oncologist will discuss the study with the patient and family.
Sampling Method: Non-Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2016-08-25 (Actual); Primary Completion 2019-04-17 (Actual); Study Completion 2019-04-17 (Actual)

PRIMARY OUTCOMES:
Early gastrointestinal toxicity | determined at 3 months
  Common Terminology Criteria for Adverse Events (CTCAE v4.0)
Late gastrointestinal toxicity | determined at 12 months
  Common Terminology Criteria for Adverse Events (CTCAE v4.0)
Early genitourinary toxicity | determined at 3 months
  Common Terminology Criteria for Adverse Events (CTCAE v4.0)
Late genitourinary toxicity | determined at 12 months
  Common Terminology Criteria for Adverse Events (CTCAE v4.0)
Early quality of life (QoL) | determined at 3 months
  EORTC QoL core questionnaire (QLQ-C30)
Early prostate specific quality of life (QoL) | determined at 3 months
  EORTC QLQ-PR25
Late quality of life (QoL) | determined at 12 months
  EORTC QoL core questionnaire (QLQ-C30)
Late prostate specific quality of life (QoL) | determined at 12 months
  EORTC QLQ-PR25

CONTACTS AND LOCATIONS:
Overall Officials: Anna Bruynzeel, MD, PhD, Principal Investigator — Amsterdam UMC, location VUmc
Locations (1):
- VU University medical center, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tetar SU, Bruynzeel AME, Oei SS, Senan S, Fraikin T, Slotman BJ, Moorselaar RJAV, Lagerwaard FJ. Magnetic Resonance-guided Stereotactic Radiotherapy for Localized Prostate Cancer: Final Results on Patient-reported Outcomes of a Prospective Phase 2 Study. Eur Urol Oncol. 2021 Aug;4(4):628-634. doi: 10.1016/j.euo.2020.05.007. Epub 2020 Jun 12. PMID 32536573